CLINICAL TRIAL: NCT05385068
Title: An Open-label, Single-arm, Phase II Study to Investigate the Efficacy and Safety of Niraparib Combined With Anlotinib Maintenance Retreatment in PSR Ovarian Cancer Patients, Who Have Previously Received PARPi Maintenance Treatment.
Brief Title: A Phase II Trial to Explore Niraparib and Anlotinib Maintenance Retreatment in Platinum-Sensitive Recurrent Ovarian Cancer Patients Previously Treated With PARPi
Acronym: t
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL2306-921
Record Dates: First submitted 2022-05-11; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Platinum-Sensitive Recurrent Ovarian Cancer; maintanence retreatment; niraparib combined with anlotinib
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — niraparib; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib combined with Anlotinib (Experimental): Participants received Niraparib 200mg or 300mg QD PO continually and Anlotinib 10mg QD PO on Days 1-14 (21 days/cycle) .
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib 200 or 300mg* QD PO continually;
  *The starting dose of niraparib was individualized based on patients' bodyweight and baseline platelet count; 200 mg QD for Patients with baseline body weight <77 kg or platelets count <150,000/μL;300 mg QD for Patients with baseline body weight ≥77 kg and platelets count ≥150,000/μL.
  For patients who had experienced grade 4 adverse events from previous use of PARPi, niraparib staring dose was 200 mg QD.
  Anlotinib 10mg QD PO from Day 1 to 14 of every 21-day cycle
  Other Names: Anlotinib

SUMMARY:
This study will be an open-label, single-arm, prospective, exploratory phase II trial to investigate the efficacy and safety of niraparib maintenance retreatment in platinum- sensitive recurrent (PSR) epithelial ovarian cancer (EOC) patients (including patients with primary peritoneal and/or fallopian tube cancer).

DETAILED DESCRIPTION:
This study will investigate the efficacy and safety of niraparib maintenance re-treatment in patients with PSR non-mucinous EOC, who have previously received maintenance therapy with a Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerisation inhibitor (PARPi) and a complete or partial radiological response to subsequent treatment with platinum-based chemotherapy or may have no evidence of disease (if optimal cytoreductive surgery was conducted prior to chemotherapy). Patients will be enrolled, given niraparib and anlotinib maintenance treatment until disease progression or untolerated toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Female patients ≥18 years of age, with histologically diagnosed platinum sensitive recurrent high-grade serous or endometrioid epithelial ovarian cancer (EOC) (including primary peritoneal and/or fallopian tube cancer).
* BRCA mutation status is known.
* Patients must have received one prior PARPi therapy, PARPi therapy includes any agent (including niraparib) used in a maintenance setting and the duration of maintenance treatment ≥6 months.
* Patients had received ≤3 lines of chemotherapy, the time between the penultimate line of platinum-containing chemotherapy and the last platinum-containing chemotherapy was > 6 months. For example, if a patient receives a non-platinum type of chemotherapy between the penultimate line of platinum-containing chemotherapy and the last platinum-containing chemotherapy, patient will be eligible if all the eligibility criteria are met.
* The most recent round of platinum-containing chemotherapy should have included ≥4 cycles of treatment , in the opinion of the investigator, in response (partial or complete radiological response) or may have no evidence of disease (if optimal cytoreductive surgery was conducted prior to chemotherapy) .
* Patients must have either CA-125 in the normal range or CA-125 decrease by more than 90% during last line chemotherapy and that is stable for at least 7 days (ie, no increase > 15% from nadir).
* Patients can have received bevacizumab during this course of treatment. Bevacizumab use as part of an earlier line of therapy is permitted.
* Patients must be enrolled within 8 weeks of their last dose of chemotherapy (last dose is the day of the last infusion).
* Patients must have a life expectancy ≥4 months.
* Eastern Cooperative Oncology Group performance status 0-2.
* Patients must have normal organ and bone marrow function, defined as follows: Absolute neutrophil count ≥ 1,500/μL; Platelets ≥ 100,000/μL; Hemoglobin ≥ 10 g/dL; Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault equation; Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN; Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Negative serum or urine pregnancy test prior to receiving the first dose of study treatment and willing to use adequate contraception to prevent pregnancy or must agree to abstain from heterosexual activity throughout the study, starting with enrollment through 90 days after the last dose of study treatment; or women of with no potential fertility.
* Ability to comply with protocol.
* All of the adverse events caused by chemotherapy recovered to Common Terminology Criteria Adverse Events (CTCAE) grade 1 or baseline, except for stable sensory neuropathy or hair loss ≤ CTCAE grade 2.

Exclusion Criteria:

* Allergy to active or inactive ingredients of niraparib or drugs with similar chemical structures.
* Allergy to active or inactive ingredients of anlotinib or drugs with similar chemical structures.
* Active and uncontrollable brain metastasis or leptomeningeal metastasis. Patients with spinal cord compression can still be considered if they have received targeted treatment and have evidence of clinical stability of the disease for at least > 28 days (controlled brain metastasis must have received radiotherapy or chemotherapy at least 1 month prior to study entry; patients may not have new symptoms related to brain lesions or symptoms indicating disease progression and either take stable dose of hormone or do not need to take hormone).
* Major surgery performed within 3 weeks before enrollment, or any surgical effects that have not recovered from the surgery, or chemotherapy.
* Palliative radiotherapy encompassing >20% of the bone marrow within 1 week of the first dose of study treatment.
* Any other malignant tumor exclude ovarian cancer has been diagnosed within 2 years before enrollment (except for completely treated basal or squamous cell skin cancer).
* Current or previous myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML).
* Other severe or uncontrolled diseases, including but not limited to: Uncontrollable nausea and vomiting, inability to swallow study drug, and any gastrointestinal disease that may interfere with the absorption and metabolism of the drug; Active viral infections, such as human immunodeficiency virus, hepatitis B virus, hepatitis C virus and so on; Uncontrolled epileptic seizures, unstable spinal cord compression, superior vena cava syndrome or other psychiatric disorders that may affect patients' informed consent; Immunodeficiency (except for splenectomy), or other diseases that investigators believe may expose patients to high-risk toxicity.
* Have the risk or tendency of bleeding and history of thrombosis: CTCAE grade 2 bleeding event occurred within 3 months prior to screening or CTCAE ≥ grade 3 bleeding event occurred within 3 months prior to screening;
* Have history of gastrointestinal bleeding or confirmed bleeding tendency within 6 months prior to screening. e.g. esophageal varices with bleeding risk, local active ulcer focus or fecal occult blood above ++.
* Have active bleeding or coagulation dysfunction, have bleeding risk or undergoing thrombolytic or anticoagulant therapy: Need anticoagulant therapy with warfarin or heparin; Need long-term anti-platelet therapy (e.g. aspirin, clopidogrel)
* Have occurred thrombus or embolism event in past 6 months, e.g. cerebral vascular accident（including transient cerebral ischemic attack), pulmonary embolism.
* A history of severe cardiovascular disease: New York Heart Association (NYHA) grade 3/4 congestive heart failure (CHF); Unstable angina or newly diagnosed angina/myocardial infarction within 12 months prior to screening; Cardiac arrhythmia despite need medication (patients taking β-receptor blockers or digoxin can be enrolled); CTCAE ≥ grade 2 valvular heart disease; Poorly controlled hypertension (systolic pressure>150 mmHg or diastolic pressure>100 mmHg)
* The following laboratory indexed are abnormal: Hyponatremia (serum sodium < 130 mmol/L); baseline serum potassium < 3.5 mmol/L (potassium supplements can be used to restore serum potassium above this before enrollment);Thyroid dysfunction and cannot maintain normal despite medical treatment
* Previous/current diseases and treatment or abnormal laboratory indexed those interfere with study result or participation of the whole study; or the investigator confirmed not suitable for this trial; have platelet or red blood cell transfusion within 4 weeks prior to the first dose of study treatment.
* Patients must not be pregnant, breastfeeding, or expecting to conceive children, while receiving study treatment.
* Corrected QT interval（QTc>450 milliseconds); if patients have QTc prolongation because of cardiac pacemaker confirmed by investigator and no other cardiac disorder, whether enrollment need further discussion with investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 1 year
  PFS is assessed as the time from niraparib treatment initiation to the earlier date of assessment of progression, as assessed by RECIST v1.1 criteria based on Investigator assessment, or death by any cause in the absence of progression

SECONDARY OUTCOMES:
Progression Free Survival (PFS) Rate at 6 months | 6 months
  PFS rate at 6 months is defined as the proportion of participants who have not progressed or died within 6 months after niraparib treatment initiation. Progression will be assessed by RECIST v1.1 criteria per investigator assessment）
Time to First Subsequent Therapy (TFST) | The date of initiation of niraparib treatment in the current study to the start date of the first subsequent anticancer therapy assessed up to 15 months.
  TFST is defined as the date of initiation of niraparib treatment in the current study to the start date of the first subsequent anticancer therapy.
Overall Survival (OS) | From the time of enrollment to date of death by any cause assessed up to 36 months.
  OS is defined as the date of initiation of niraparib treatment to the date of death by any cause.
Frequency and severity of adverse effects as defined by CTCAE version 5.0 | From the time of enrollment to date of 30 days after the last study drug administration.
  Number of patients with any non-serious adverse event (non-SAE) or any SAE to evaluate the safety and tolerability of niraparib combined with anlotinib.